CLINICAL TRIAL: NCT06397144
Title: A PHASE 1, OPEN-LABEL, RANDOMIZED, SINGLE DOSE, CROSSOVER STUDY TO DETERMINE THE BE OF NIRMATRELVIR FOLLOWING ORAL ADMINISTRATION OF FDC TABLETS RELATIVE TO THE PAXLOVID® COMMERCIAL TABLETS IN HEALTHY ADULT PARTICIPANTS UNDER FASTED CONDITIONS
Brief Title: A Study on 2 Different Combination Tablets of Nirmatrelvir Plus Ritonavir to Compare Them With Marketed Paxlovid in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor business decision to terminate study. Decision not due to major safety concerns or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671009; NCT06397144 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Biological Availability; Healthy Participants
Keywords: Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Nirmatrelvir; Paxlovid
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination; nirmatrelvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Paxlovid commercial tablets A (Low Dose) (Active Comparator): Single oral dose of nirmatrelvir/ ritonavir 150 (1 × 150)/100 mg commercial tablets under fasted conditions (Reference 1)
  Interventions: Drug: Paxlovid
- Paxlovid commercial tablets B (High Dose) (Active Comparator): Single oral dose of nirmatrelvir/ ritonavir 300 (2 × 150)/100 mg commercial tablets under fasted conditions (Reference 2)
  Interventions: Drug: Paxlovid
- Nirmatrelvir/ritonavir FDC tablets Test formulation 1 (Experimental): Single oral dose of nirmatrelvir /ritonavir 150/100 mg (2 × [75/50 mg]) FDC tablets Test formulation 1 (Test 1)
  Interventions: Drug: Nirmatrelvir/ritonavir
- Nirmatrelvir/ritonavir FDC tablets Test formulation 2 (Experimental): Single oral dose of nirmatrelvir/ ritonavir 300/100 mg (2 × [150/50 mg]) FDC tablets Test formulation 2 (Test 2)
  Interventions: Drug: Nirmatrelvir/ritonavir

INTERVENTIONS:
Drug: Paxlovid — Reference 1
  Other Names: Nirmatrelvir/ritonavir commercial tablets
  Arms: Paxlovid commercial tablets A (Low Dose)
Drug: Paxlovid — Reference 2
  Other Names: Nirmatrelvir/ritonavir commercial tablets
  Arms: Paxlovid commercial tablets B (High Dose)
Drug: Nirmatrelvir/ritonavir — Test 1
  Other Names: Nirmatrelvir/ritonavir FDC test tablets formulation 1
  Arms: Nirmatrelvir/ritonavir FDC tablets Test formulation 1
Drug: Nirmatrelvir/ritonavir — Test 2
  Other Names: Nirmatrelvir/ritonavir FDC test tablets formulation 2
  Arms: Nirmatrelvir/ritonavir FDC tablets Test formulation 2

SUMMARY:
Medicines that may have different names or be made in different ways but have the same effect on the body are called bioequivalent.

The purpose of this study is to learn about the bioequivalence of nirmatrelvir plus ritonavir after taking 2 different combination tablet forms by mouth. These combination tablets are compared to the tablet formulation that is already in the market. This study will be done under fasted conditions in healthy adult participants.

This study is seeking participants who are:

* Male and non-pregnant female participants aged 18 years and above.
* with a body weight of more than 50 kilograms and Body Mass Index (BMI) between 16 to 32 kilograms per meter squared.
* are healthy as confirmed by medical history, physical examination, laboratory tests.

The study will also look at the safety and tolerability of nirmatrelvir plus ritonavir combination tablet and marketed tablet formulations in healthy adult participants.

The study will consist of 4 treatments:

Treatment A: Single oral dose of nirmatrelvir plus ritonavir 150 (1 × 150)/100 milligrams marketed tablets under fasted conditions (Reference 1) Treatment B (low dose strength): Single oral dose of nirmatrelvir plus ritonavir 150/100 milligrams (2 × [75/50 milligrams]) combination tablets under fasted conditions (Test 1) Treatment C: Single oral dose of nirmatrelvir/ritonavir 300 (2 × 150)/100 milligrams marketed tablets under fasted conditions (Reference 2) Treatment D (high dose strength): Single oral dose of nirmatrelvir/ritonavir 300/100 milligrams (2 × [150/50 milligrams]) combination tablets under fasted conditions (Test 2)

All treatments will be given under fasted conditions. Fasted condition means the participants would not have had anything to eat before taking the medicines.

Around 28 participants will be enrolled in the study. Healthy participants will be tested to see if they can be in the study within 28 days before receiving the study medicine. Selected participants will be admitted to the clinical research unit (CRU) one day before receiving the study medicine and will remain in the CRU until discharge after completing all the treatment periods.

On Day 1 of each period, participants will be given a single dose of study medicine nirmatrelvir/ritonavir 300/100 mg or 150/100 mg by mouth by chance. Study medicine will be given with approximately 240 milliliters of room temperature water under fasted conditions (overnight fast of at least 10 hours and no food until 4 hours after receiving the study medicine). Blood samples will be collected at different times of the day up to 48 hours after taking the study medicine. Participants will be discharged from the CRU on Day 3 of Period 4, after all the study related procedures have been completed.

A follow-up call will be made to participants around 28 to 35 days from receiving the final dose of the study medicine. The study will look at the experiences of participants receiving the study medicine. This will help to understand if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and standard 12-lead ECG (electrocardiogram).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Female participants of childbearing potential must have a negative pregnancy test at screening and on Day -1.
* BMI (Body Mass Index) of 16-32 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD (Informed consent Document) and in this protocol.

Exclusion Criteria:

* Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of HIV (Human Immunodeficiency Virus) infection, Hepatitis B, or Hepatitis C; positive testing for HIV, HBsAg (Hepatitis B surface Antigen), HBcAb (Hepatitis B core Antibody) or HCVAb (Hepatitis C Virus Antibody). Hepatitis B vaccination is allowed.
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Participants who have received a COVID-19 vaccine within 7 days before screening or admission, or who are to be vaccinated with a COVID-19 vaccine at any time during the study confinement period.
* A positive urine drug test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Area under curve (AUC) from time zero to 48 hours post dose (nirmatrelvir) | 0 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours
Peak plasma concentration (Cmax) for nirmatrelvir | 0 , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours

SECONDARY OUTCOMES:
AUC from time zero to 48 hours post dose (ritonavir) | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours
Cmax for ritonavir | 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 and 48 hours
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 28 days after last dose of study medication
Number of Participants With Clinically Notable Vital Signs | Baseline (Day 0) up to day 3 of treatment period 4
Number of Participants With Clinically Notable Changes in Clinical laboratory results | Baseline (Day 0) up to day 3 of treatment period 4
Number of Participants With Clinically Notable Abnormality in physical examination | Baseline (Day 0) up to day 3 of treatment period 4

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671009